CLINICAL TRIAL: NCT00432302
Title: Investigation of Mass Balance and Major Metabolites After Administration of 28 mg Radiolabeled ZK 219477 in Patients With Solid Tumor in an Open-label, Non Randomized Design
Brief Title: Investigation of Mass Balance of the Test Drug and Major Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91490; 2006-000188-26 (EudraCT Number); 310301 (Other: Company Internal)
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms
Keywords: Cancer; Tumor; Malignancy; Mass Balance; Chemotherapy; Drug; Cancer Treatment; Intravenous Infusion; Epothilone; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sagopilone (Experimental): Subjects received 28 mg ZK 219477, containing 14 kBq/7.8 µg [14C]-ZK 219477 in the first infusion (Treatment course 1) followed by subsequent infusions (Treatment courses 2 to n [till disease progression]) of 16 mg/m2 ZK 219477 without radioactive label. Interval between the treatments was at least 21 days.
  Interventions: Drug: Sagopilone (BAY 86-5302, ZK 219477)

INTERVENTIONS:
Drug: Sagopilone (BAY 86-5302, ZK 219477) — First infusion only: 28 mg, containing 14 kBq/7.8 mcg [14C]-ZK 219477. Subsequent infusions: 16 mg/m2 ZK 219477 without radioactive label. IV infusion was given over a period of 30 min.

SUMMARY:
The purpose of this study is to: a) Determine how the body takes up the test drug and distributes it into various body organs and tissues, how it processes the drug and how it ultimately removes it; and b) Examine how well the test drug works against cancer, and whether it is safe and tolerable to take

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years; female ≥ 50 years without childbearing potential (confirmed by either: age ≥ 60; or history of hysterectomy; or hormone analysis in serum: Estradiol ≤ 20 pg/mL and follicle stimulating hormone ≥ 40 IU/L)
* Solid tumor
* Adequate function of major organs
* Failed previous cancer treatment
* Peripheral venous access

Exclusion Criteria:

* Concurrent severe and/or uncontrolled disease
* Brain tumors
* Marked constipation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Blood, urine and fecal samples will be collected over a period of 336 hours (14 days) to measure 14C, ZK 219477 and its major metabolites following the intravenous administration of 14C-ZK 219477. | 14 days
Cmax | 14 days
  Maximum plasma concentration for [14C]-ZK 219477, ZK 219477
tmax | 14 days
  Time to Cmax for [14C]-ZK 219477, ZK 219477
AUC | 14 days
  Area under the concentration time curve for [14C]-ZK 219477, ZK 219477
AUC(0-tlast) | 14 days
  AUC from administration until the last time point with measurable concentration for [14C]-ZK 219477, ZK 219477
AUC(0-24) | 14 days
  AUC from time zero to 24 hours for [14C]-ZK 219477, ZK 219477
MRT | 14 days
  Mean residence time for [14C]-ZK 219477, ZK 219477
t1/2 | 14 days
  Terminal half-life for [14C]-ZK 219477, ZK 219477
λz | 14 days
  Apparent terminal rate constant for [14C]-ZK 219477, ZK 219477
CL | 14 days
  Total clearance for ZK 219477
Vss | 14 days
  Apparent volume of distribution at steady state for ZK 219477
Vz | 14 days
  Apparent volume of distribution during terminal phase for ZK 219477

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 12 weeks to 30 weeks
Overall response | Approximately 10 to 32 weeks
  Determination of complete response (CR), partial response (PR), unknown, stable disease, progressive disease (PD) by the modified Response Evaluation Criteria in Solid Tumors
Best overall response | Approximately 10 to 32 weeks
  Overall response as obtained at all time points available for an individual subject combined to the 'best overall response'
Responders | Approximately 10 to 32 weeks
  'Response' was considered to be established if 'Best overall response' of PR or CR was confirmed at any time after the start of study treatment. If response was established, a subject was referred to as a 'responder'

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Liège, Belgium

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/